CLINICAL TRIAL: NCT03768778
Title: Non-Missile Penetrating Brain Injuries, Cases Registry in Sohag University Hospital
Brief Title: Non-missile Penetrating Head Trauma,Cases Registry in Sohag University Hospital
Acronym: trauma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, ahmed salaheldin mohammed saro, Assistant professor of neurosurgery, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Sohag1
Record Dates: First submitted 2018-12-04; First posted 2018-12-07 (Actual); Last update posted 2018-12-10 (Actual); Status verified 2018-12

CONDITIONS: Head Injuries With Non Missile Penetrating Objjects
Keywords: Penetrating brain trauma (PBT),Traumatic brain injury (TBI), Intensive care unit, non missile.
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Debridement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Debridement (Other)
  Interventions: Procedure: Debridement and dural repair

INTERVENTIONS:
Procedure: Debridement and dural repair
  Other Names: Removal of foreign bodies with dural and vascular repair

SUMMARY:
A retrospective study was done in Neurosurgery trauma unit, Sohag University. Eighteen patients reported with different mechanisms of trauma. All patients clinically tested involving neurological evaluation. Computed tomography brain was done for them at the time of admission. Cautious removal of the penetrating object with local debridement of surrounding tissues including skin, skull, dura and brain tissue and watertight closure of the dura should be done. Patients transferred to the Intensive care unit (ICU) for 48 - 72 hours.

DETAILED DESCRIPTION:
Traumatic intracranial penetration of foreign non-missile object rarely occurs. Early mortality may be caused by hemorrhages, major vascular injury or contusions; while epileptic seizures and infections are among the possible complications in later stages. Complete excision of the foreign object should be done for all patients and any dural and/or vascular injuries should be repaired during surgical treatment.

Neurological level, hemodynamic and respiratory status at hospital admission, type of penetrating the object, pupil size, and reactivity, as the CT findings, all these factors will affect the prognosis so they should be evaluated carefully before the decision of the line of management. Intracranial infection, CSF leak and recurrent attacks of convulsions are the most common complications.

Our goal in this study to report cases with non-missile penetrating head injuries and evaluate the possible predictive factors in a series of 18 patients sustaining penetrating head injuries, admitted to our hospital over a period of 2 years, to be used as a guide for the surgical management.

ELIGIBILITY:
Inclusion Criteria:

* Any patient with penetrating head trauma

Exclusion Criteria:

* missile penetrating head injuries

Ages: 4 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 18 (Actual)
Dates: Start 2012-11-01 (Actual); Primary Completion 2014-10-01 (Actual); Study Completion 2014-10-01 (Actual)

PRIMARY OUTCOMES:
(Glasgow Coma Scale)(GCS) to evaluate non-Missile Penetrating Brain Injuries | 2 years
  Descriptive scale grades from (3 to 15). 3 is worst and 15 is the best

IPD SHARING:
Plan to Share IPD: Undecided